CLINICAL TRIAL: NCT04874220
Title: Neural Correlates of Real World Spatial Navigation in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nanthia Suthana, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-001459
Record Dates: First submitted 2021-04-28; First posted 2021-05-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Memory, Delayed
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep brain stimulation will be used

SUMMARY:
The purpose of this study is to understand the neural mechanisms that support real world spatial navigation in humans using deep brain recordings and stimulation during virtual reality (VR), augmented reality, and real world memory tasks. We will determine the cognitive (i.e., memory) and behavioral (i.e., body, head, eye position and movement) factors that modulate deep brain activity and the consequent effects of memory-enhancing deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older and has undergone RNS system placement
* Willing to provide informed consent and participate the study
* Ability to read and write English fluently

Exclusion Criteria:

* Unwilling to provide informed consent

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Spatial memory | Throughout study completion, an average of 2-4 days per year
  Spatial memory will be measured using virtual, augmented and real-world spatial navigation tasks where participants will be asked to navigate a previously learned rout as well as if they recognize objects (i.e. landmarks) that appeared along the route (photos of seen landmarks vs unseen landmarks).
Memory performance change | Throughout study completion, an average of 2-4 days per year
  Memory performance will be measured using excess path length, latency, and accuracy rate.
Oscillatory activity change | Throughout study completion, an average of 2-4 days per year
  Changes in theta, gamma, and theta-gamma coupling will be measured both in relation to changes in memory performance on trials with and without deep brain stimulation as well as in relation to body, head, and eye position in a virtual, augmented, or real-world environment.

CONTACTS AND LOCATIONS:
Overall Officials: Nanthia Suthana, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data collected for this research represent a valuable resource to the scientific community, and the PIs will make them accessible to others, while respecting the special needs for confidentiality. All data will be anonymized before being provided to the scientific community. Researchers can also request access to the data under collaborative and co-authorship agreements prior to the end of the funding period or before publication. The results from the proposed project will also be shared at scientific meetings (local, national and international) as well via published manuscripts.
Time Frame: All data will be provided by the time publication occurs or when the proposed funding period has ended.
Access Criteria: Researchers can request access to the data under collaborative and co-authorship agreements prior to the end of the funding period or before publication.